CLINICAL TRIAL: NCT04647331
Title: Betalactam Pharmacokinetics in Endocarditis Patients
Status: Recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02886
Record Dates: First submitted 2020-11-19; First posted 2020-11-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-09

CONDITIONS: Infective Endocarditis
Keywords: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infectious endocarditis (IE) is associated with mortality rates of 10-12%. Adequate antibiotic therapy is crucial for survival and is administered in high doses due to the severity of the disease. In most cases, beta-lactam antibiotics (e.g. ampicillin, penicillin G, cefotaxime or cloxacillin) are employed. A number of patient characteristics, such as age, body weight, and renal function) influence the pharmacokinetics of these drugs. Yet, the interindividual variability is poorly understood meaning that a large proportion of patients are at risk of subtherapeutic or excessive drug concentrations that might result in treatment failure or side effects, respectively.

In the present study, data will be collected on antibiotic concentrations in patients treated with beta-lactams for infectious endocarditis as well as patient characteristics and treatment outcomes. A mathematical model will be developed to determine which patient factors determine drug pharmacokinetics. Based on this model, predictions will be made by mathematical simulations on which dosing regimens are optimal for individual patients to ensure therapeutic and non-toxic drug concentrations. In total, 150 patients will be included at four University Hospitals in Sweden; Uppsala University Hospital, Sahlgrenska University Hospital in Gothenburg, Skåne University Hospital in Lund and Karolinska University Hospital in Stockholm. Following informed consent to participate blood samples will be collected at 6 time-points during a dose interval and then at 3 time-points weekly during the full treatment episode (maximum 6 weeks).

DETAILED DESCRIPTION:
Objectives The primary objective of the study is to determine the pharmacokinetics of beta-lactam antibiotics in patients with infectious endocarditis, and how the pharmacokinetic profile is associated with various patient factors (e.g. age, body weight, renal function). Secondary objectives are to descriptively assess potential associations between drug exposure, pharmacokinetic/pharmacodynamic targets and clinical outcomes.

Inclusion of patients and sample size Patients are prospectively included at the departments of infectious diseases, internal and acute medicine, cardiology and thoracic surgery at four University Hospitals in Sweden; Uppsala University Hospital, Sahlgrenska University Hospital in Gothenburg, Skåne University Hospital in Lund and Karolinska University Hospital in Stockholm. Potential participants are screened for using the electronic medical records. Inclusion criteria are as follows: (1) admission at one of the study wards, (2) a diagnosis of probable or verified infectious endocarditis, (3) treatment with ampicillin, penicillin G, cefotaxime or cloxacillin and (4) informed written consent to participate in the study. The following exclusion criteria will be applied: (1) age less than 18 years and (2) ongoing or planned hemodialysis.

Based on previous research using similar methods, 30 patients per antibiotic substance (total 150 patients) is considered sufficient to develop a robust mathematical model.

Collection of blood samples and patient data Following inclusion, a series of samples will be taken within one week from start of treatment. Beta-lactams are normally prescribed at 6-8 h dose intervals. One series of 6 blood samples will be collected at 0, 0,5, 1, 2, 4 and 6 or 8 h (depending on dose interval, prior to next dose) after administration of antibiotics. Thereafter, samples will be collected once weekly and 0, 3 or 4 (mid-dose interval) and 6 or 8 h (depending on dose interval, prior to next dose).

Information on patient characteristics, including age, body weight, and gender, will be obtained from the electronic medical records. Further, the results of biomarkers (e.g. albumin, creatinine, CRP), collected as part of routine practice, will be noted. If not collected as standard of care, patients will be subject to extra samples to ensure biomarkers are monitored at least twice weekly.

Clinical outcomes Treatment failure is defined as mortality during antibiotic treatment for infectious endocarditis or relapse of endocarditis within 6 months after completion of therapy with isolation of the same pathogens as in the initial episode. Other indicators of treatment failure include acute surgery for endocarditis, clinical deterioration resulting in transfer to the ICU, thromboembolic events more than 7 days after initiation of antibiotics and resistance development of the causative bacteria. The following side effects will be monitored: deterioration of renal impairment, allergic reaction suspected to be caused by the antibiotic treatment, Clostridioides difficile enteritis or other suspected side effects resulting in a shift of therapy to another antibiotic.

Handling of samples and data Blood samples will be stored at -70 degrees Celsius at the Department of infectious diseases at the respective hospital where the samples have been collected. The samples will be sent to Sahlgrenska University Hospital, Gothenburg, for determination of drug concentrations.

Patient names and personal identification numbers will be replaced by a number. Personal data will be stored at the Department of infectious diseases at the respective hospital where the patient has been included. Only the responsible researchers will have access to the code key and be able to link personal information to the individual participants. All information will be handled in accordance with the General Data Protection Regulation (GDPR) and all analyses and presentation of data will be performed using anonymous data.

Mathematical modeling and simulations The collected drug concentrations will be analyzed by non-linear mixed effects modeling using NONMEM. Associations between administered dose and the measured drug concentration over time will be described (pharmacokinetics). Correlations with patient characteristics and biomarkers, as well as clinical outcomes in terms of cure, mortality and documented side effects (pharmacodynamics) will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Verified or suspected left or right sided endocarditis in native or prosthetic valve
* Intravenous antibiotic therapy with either ampicillin, penicillin G, cefotaxime or cloxacillin
* Signed informed consent to participate in study

Exclusion Criteria:

* <18 years of age
* Ongoing dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients in Uppsala University Hospital treated for verified or suspected left or right sided endocarditis in nativ or prosthetic valve with intravenous antibiotic therapy (ampicillin, cefotaxime, cloxacillin or penicillin G).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Determinants of the pharmacokinetic profiles of betalactam antibiotics ampicillin, cefotaxime, cloxacillin and penicillin G | 6 years
  Data on drug concentrations will be analysed using non-linear mixed effect modeling to describe correlations between the observed concentrations and the administered dose, patient characteristics (e.g., age, body weight, gender) or biomarkers (e.g. albumin, creatinine, CRP)
Maximum drug concentration (Cmax) of betalactam antibiotics ampicillin, cefotaxime, cloxacillin and penicillin G | 6 years
  Data on drug concentrations will be analysed using non-linear mixed effect modeling to determine Cmax.
Volume of distribution (Vd) of betalactam antibiotics ampicillin, cefotaxime, cloxacillin and penicillin G | 6 years
  Data on drug concentrations will be analysed using non-linear mixed effect modeling to determine Vd.
Clearance (CL) of betalactam antibiotics ampicillin, cefotaxime, cloxacillin and penicillin G | 6 years
  Data on drug concentrations will be analysed using non-linear mixed effect modeling to determine CL.
Half-life (t1/2) of betalactam antibiotics ampicillin, cefotaxime, cloxacillin and penicillin G | 6 years
  Data on drug concentrations will be analysed using non-linear mixed effect modeling to determine t1/2.
Time above the minimum inhibitory concentration (T>MIC) of betalactam antibiotics ampicillin, cefotaxime, cloxacillin and penicillin G | 6 years
  Data on drug concentrations will be analysed using non-linear mixed effect modeling to determine T>MIC.
Area under the curve (AUC) of betalactam antibiotics ampicillin, cefotaxime, cloxacillin and penicillin G | 6 years
  Data on drug concentrations will be analysed using non-linear mixed effect modeling to determine AUC.

SECONDARY OUTCOMES:
Mortality | 12 months
  All cause mortality
Remission of disease | 12 months
  Relapse in infective endocarditis within 6 months
Thromboembolic event | 12 months
  Stroke or embolic event related to endocarditis
Resistance development | 12 months
  Resistance development in causing pathogen during treatment assessed with repeated blood culture samples for assessment of bacterial growth and antibiotic susceptibility testing
Renal failure | 12 months
  Elevation of creatinine clearance of at least 30% during antibiotic treatment
Clostridioides difficile infection | 12 months
  Positive culture of C. difficile during and within 6 months of discontinued antibiotic treatment
Adverse events | 12 months
  Adverse events related to antimicrobial therapy
Associations between antibiotic pharmacokinetics and outcome | 12 months
  Potential associations between suboptimal antibiotic concentrations, in relation to established pharmacokinetic/pharmacodynamic targets, and any of the secondary outcomes will be described (exploratory)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Tängdén, MD, Phd, Principal Investigator — Uppsala University Hospital
Locations (4):
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Lund
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: No